CLINICAL TRIAL: NCT02054299
Title: Effects of Genetic Polymorphisms in the Organic Cation Transporter OCT1 on Cellular Uptake and Metabolism of Antidepressants and Other Organic Cationic Drugs
Brief Title: Open Label Pharmacokinetic-Pharmacogenetic Study on Polymorphisms in the Organic Cation Transporter OCT1
Acronym: PG-OCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Johannes Matthaei, Sub-investigator, Principal investigator is Prof. Juergen Brockmoeller, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PG-OCT; 2012-003546-33 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Drug Metabolism; Membrane Transport

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug application (Experimental): 6 treatment periods. On each period one of the following interventions
  Interventions: Drug: Drug application Amitriptyline; Drug: Drug application Desvenlafaxine; Drug: Drug application Sumatriptan; Drug: Drug application Proguanil; Drug: Drug application Fenoterol; Drug: Drug application Thiamine

INTERVENTIONS:
Drug: Drug application Amitriptyline — Amitriptyline: 25 mg, single oral application
Drug: Drug application Desvenlafaxine — Desvenlafaxine: 50 mg, single oral application
Drug: Drug application Sumatriptan — Sumatriptan: 50 mg, single oral application
Drug: Drug application Proguanil — Proguanil: 200mg, single oral application
Drug: Drug application Fenoterol — Fenoterol: 180 mcg, single intravenous application
Drug: Drug application Thiamine — Thiamine: 200mg, single oral application

SUMMARY:
The purpose of this study is to determine the effect of the organic cation transporter OCT1 polymorphisms on the pharmacokinetics of several drugs in order to explain efficacy and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to study entry including informed consent for molecular genetic analysis concerning candidate genes relevant for pharmacokinetics and pharmacodynamics of the study medication.
2. Both genders (male and female), as far as feasible, in each of the 3 OCT1 genotype groups, an equal proportion of males and females will be included.
3. Healthy adults aged ≥18 to < 50 years
4. Body weight not less than 48 kg and body mass index (BMI) not less than 17 kg/m² and not greater than 32 kg/m².
5. Willingness to meet the study instructions and to co-operate with the study personal
6. No clinically relevant pathological findings in any of the investigations at the screening visit. Minor deviations of laboratory values from the normal range may be accepted, if judged by the investigator to have no clinical relevance
7. Systolic blood pressure ≤ 140 mmHg and ≥ 100 mmHg, diastolic blood pressure ≤ 90 mmHg and ≥ 60 mmHg and heart rate ≤ 90 bpm and ≥ 50 bpm at screening visit
8. Female subjects will only be included if they express their willingness not to become pregnant during the entire study period by practicing abstinence or reliable methods of contraception as specified in the respective protocol section.

Exclusion Criteria:

1. Unwillingness or inability to give informed consent
2. Involvement in the planning and conduct of the study (applies to staff directly employed at the study site / department)
3. Participation in a clinical study or use of any other investigational or non-registered drug or vaccine during the study period or within 30 days preceding the first dose of study drugs.
4. Blood, plasma or thrombocyte donation during the last 15 days prior to application of the test drugs.
5. Any planned surgical treatment during the last 14 days prior and 14 days after the application of the test drugs.
6. Known pregnancy or lactation period
7. Any relevant pathological findings in any of the investigations at the screening visit including significant abnormalities as result of the medical-screening-laboratory-analysis, especially of the liver and kidney related parameters unless judged as medically irrelevant.
8. QTcF > 450 ms in screening ECG
9. Systolic blood pressure > 140 mmHg and < 100 mmHg, diastolic blood pressure > 90 mmHg and < 60 mmHg and heart rate > 90 bpm and < 50 bpm pre-dose at treatment period 4 (Amitriptyline)
10. Any disease affecting liver or kidney or impairment of the liver or kidney-function
11. Any cardiovascular disease
12. Moderate to severe hypertension requiring medication therapy
13. Bronchogenic asthma requiring constant drug treatment (stages 2 to 4 asthma)
14. Diabetes mellitus, hyperthyroidism, hypothyroidism
15. Glaucoma
16. Symptomatic prostatic hyperplasia
17. Any medical constellation that increases risk of bleeding, including chronic treatment with NSAID or COX-2 inhibitors
18. History of alcohol and/or drug abuse and/or any abusive use of medicaments and/or positive drug screen
19. History of any psychiatric or neurologic disorder. If there are any doubts at the screening visit on whether a person is suffering from a depression or not he or she will be excluded from the study or examined by a psychiatrist for clarification before inclusion.
20. Any major gastrointestinal disease and any gastrointestinal disorder that is expected to significantly interfere with the pharmacokinetics of the study drug
21. Gastrointestinal surgery which may interfere with the pharmacokinetics of the study drug (except appendectomy or herniotomy)
22. Taking any medication within 7 days before or during the trial with the following exceptions: Oral contraceptive drug used will be documented but will not be an exclusion criterion. Other medication might be allowed on single case basis if considered necessary for the subject's safety and well-being and if interactions with the study medication are judged as irrelevant.
23. Any other findings that could compromise the safety of the participant or the quality of the study-results
24. Any known hypersensitivity or allergic reactions to any of the tested drugs
25. History of severe hypersensitivity reactions and anaphylaxis
26. Any other clinically significant diseases as judged by the investigator
27. Body temperature > 37.5°C prior to drug application
28. Known infection with HIV, Hepatitis B (HBsAg) or Hepatitis C (no laboratory diagnostics concerning these diseases will be performed within the present study)
29. Inability or unwillingness to avoid any intake of alcohol from 48 h prior to until 72 hours after Investigational Medicinal Product (IMP) application application
30. Pregnancy (positive pregnancy test performed prior to drug administration)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of the investigational drugs | up to 60 hours

SECONDARY OUTCOMES:
Total clearance, Cmax, Tmax, Mean AbsorptionTime, Alpha and Beta half-lives, Mean Residence Time (MRT) and Volume of distribution of the investigated drugs and their metabolites | up to 60 hours
Dry mouth, fatigue, nausea, headache, vertigo, tinnitus, chills, anxiety and difficulties to read on Visual Analog Scales. | up to 60 hours
Sedation on Stanford sedation scale | up to 60 hours
Pupil diameter, latency, diameter at maximal constriction, amplitude and time for 33% recovery of initial pupil diameter measured by pupillometrie | up to 60 hours
Genetic variants in OCT1, CYP2C19, CYP2D6 and MAO A | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Brockmoeller, Prof., Study Director — University Medical Center Goettingen
Locations (1):
- Department of Clinical Pharmacology, University Medical Center Goettingen, Göttingen, Germany

REFERENCES:
- [Derived] Tzvetkov MV, Matthaei J, Pojar S, Faltraco F, Vogler S, Prukop T, Seitz T, Brockmoller J. Increased Systemic Exposure and Stronger Cardiovascular and Metabolic Adverse Reactions to Fenoterol in Individuals with Heritable OCT1 Deficiency. Clin Pharmacol Ther. 2018 May;103(5):868-878. doi: 10.1002/cpt.812. Epub 2017 Dec 8. PMID 28791698